CLINICAL TRIAL: NCT04350203
Title: Surgical-Site Infection After Laparoscopic Right Colectomy: A Cohort Study Comparing Intracorporeal Anastomosis in Front of Extracorporeal Anastomosis
Brief Title: Surgical-Site Infection After Laparoscopic Right Colectomy
Status: Completed | Type: Observational
Sponsor: Hospital Plató (Other)
Responsible Party: Sponsor
Other Study IDs: HPlato
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Surgical Site Infection
Keywords: Right Colectomy; Laparoscopy; Intracorporeal Anastomosis; Extracorporeal Anastomosis; Colorectal Cancer
MeSH Terms: conditions — Surgical Wound Infection; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intracorporeal Anatomosis (IA): Laparoscopic Right colectomy with intracorporeal (IA) side-to-side isoperistaltic anastomosis
  Interventions: Procedure: Laparoscopic right colectomy with intracorporeal anastomosis (IA)
- Extracorporeal Anastomosis (EA): Patients submitted to a Laparoscopic Right Colectomy with extracorporeal anastomosis (EA)
  Interventions: Procedure: Laparoscopic right colectomy with extracorporeal anastomosis (EA)

INTERVENTIONS:
Procedure: Laparoscopic right colectomy with intracorporeal anastomosis (IA) — First, the right colon dissection was completed by laparoscopy. An isoperistaltic side-to-side ileocolonic mechanical anastomosis was then performed by using a linear cutting stapler. The enterotomy used to enter the stapler was closed with a running suture (3-0 absorbable monofilament or a 3-0 barbed suture). Finally, the specimen was extracted through a Pfannenstiel mini-laparotomy (4-5 cm).
  Groups: Intracorporeal Anatomosis (IA)
Procedure: Laparoscopic right colectomy with extracorporeal anastomosis (EA) — First, the right colon was widely mobilized. A small laparotomy was performed in the mid/upper abdomen to exteriorize the colon and to perform a side-to-side mechanical anastomosis, using a linear cutting stapler (GIA). The bowel opening was closed either with a manual suture or by a second firing of the GIA.
  Groups: Extracorporeal Anastomosis (EA)

SUMMARY:
Laparoscopic right colectomy with intracorporeal anastomosis seems to be associated with several short-term benefits. It could reduce the postoperative infection rate and shorten the hospital stay.

This study aimed to evaluate the postoperative surgical site infection (SSI) rate after laparoscopic right hemicolectomy with intracorporeal anastomosis, compared to extracorporeal anastomoses.

DETAILED DESCRIPTION:
This is a comparative cohort study of two anastomosis techniques for laparoscopic right hemicolectomy.

Between 2011 and 2019, all unselected consecutive patients who underwent a laparoscopic resection of the right colon were considered to be included in the study. The inclusion and exclusion criteria are detailed in the section below. Data were extracted from a prospectively maintained colorectal surgery database of a university-affiliated hospital in Barcelona.

All included patients signed a standard consent form after being informed about the characteristics of the procedure. Institutional board approval was obtained before the review of the patients' data.

Patients were divided into two groups, depending on the anastomotic technique performed: intracorporeal (IA) or extracorporeal.

The primary endpoint of the study was to determine the surgical-site infection (SSI) rate and its potential impact on the length of hospital stay. Anastomotic leak was defined as a "leak of luminal contents from a surgical join between two hollow viscera" according to the Surgical Infection Study Group [1]. The evaluation of SSI, intraabdominal abscess and wound infection (both superficial and deep), was based on the Centers for Disease and Prevention definitions [2].

Secondary endpoints included other short-term postoperative complications (30 days), besides the SSI: hemorrhage (intraabdominal and anastomotic), ileus (intolerance to oral feeding beyond the fourth postoperative day or the need for insertion of a nasogastric tube), evisceration, medical complications, reoperations, and mortality. The severity of the complications was reported using the Clavien-Dindo classification [3].

The following variables were also collected: operating time (from the start of the incision to skin closure), concomitant surgery performed, assistance incision site (for anastomosis or specimen retrieval), conversion rate to open surgery (need for a laparotomy wider than 10 cm.), and oncological parameters as the size of the tumor, the depth of wall invasion (T) and the lymph node harvest.

Patient demographics characteristics analyzed were age, sex, body mass index (BMI), and associated comorbidities. The anesthetic risk was measured according to the American Society of Anesthesiologists (ASA) classification system [4].

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years candidates for scheduled surgery with curative intention to resect a benign or malignant neoplasm of the right colon

Exclusion Criteria:

* stage IV disease (distant metastatic or intraabdominal disseminated disease that contraindicates surgery with curative intention)
* emergency operation for complicated disease
* medical contraindication for general anesthesia
* pregnancy
* chronic renal insufficiency requiring dialysis
* or patient refusal and/or absence of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients over 18 years candidates for scheduled surgery requiring laparoscopic right colon resection (ascendant or transverse colon)
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Anastomotic leak rate | 30 days
  percentage of clinical anastomotic leak leading to an intervention
Intraabdominal Abscess rate | 30 days
  percentage of abdominal abscess (clinical or radiological) leading to an intervention (surgical or percutaneous)
Wound Infection | 30 days
  percentage of wound infection (deep or superficial)

SECONDARY OUTCOMES:
Length of Hospital Stay | 30 days
  days that patients required hospitalization
postoperative complications 1 | 30 days
  global morbidity evaluated according the Dindo-Clavien Classification
postoperative complications 2 | 30 days
  postoperative haemorrhage needing intervention (surgical or endoscopic)
Operating time of the procedure | During the perioperative period
  Total duration of the surgical procedure (in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Hoyuela, MD, PhD, Principal Investigator — Chief, Dept. of Surgery
Locations (1):
- Hospital Plató, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peel AL, Taylor EW. Proposed definitions for the audit of postoperative infection: a discussion paper. Surgical Infection Study Group. Ann R Coll Surg Engl. 1991 Nov;73(6):385-8. PMID 1759770
- [Background] van Oostendorp S, Elfrink A, Borstlap W, Schoonmade L, Sietses C, Meijerink J, Tuynman J. Intracorporeal versus extracorporeal anastomosis in right hemicolectomy: a systematic review and meta-analysis. Surg Endosc. 2017 Jan;31(1):64-77. doi: 10.1007/s00464-016-4982-y. Epub 2016 Jun 10. PMID 27287905
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Derived] Hoyuela C, Guillaumes S, Ardid J, Hidalgo NJ, Bachero I, Trias M, Martrat A. The impact of intracorporeal anastomosis in right laparoscopic colectomy in the surgical site infections and the hospital stay: a cohort study. Updates Surg. 2021 Dec;73(6):2125-2135. doi: 10.1007/s13304-021-00998-5. Epub 2021 Feb 15. PMID 33590349
- See also: American Society of Anesthesiologists. ASA Physical Status Classification System — https://www.asahq.org/standards-and-guidelines/asa-physical-status-classification-system
- See also: Centers for Disease Control and Prevention. National Healthcare Safety Network (NHSN) Procedure-Associated (PA) Module: Surgical Site Infection (SSI) Event — http://www.cdc.gov/nhsn/PDFs/pscManual/9pscSSIcurrent.pdf